CLINICAL TRIAL: NCT03225040
Title: Cross-sectional Study of Bone Density, Bone Microarchitecture, Vertebral Fractures and Trabecular Bone Score in Patients With Acromegaly Treated With Pegvisomant Compared to Patients With Untreated Active Acromegaly
Brief Title: Bone MicroArchitecture in Acromegaly
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Pamela U. Freda, Professor of Medicine, Columbia University
Other Study IDs: AAAE5304
Record Dates: First submitted 2017-07-13; First posted 2017-07-21 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Acromegaly; Osteoporosis Risk
Keywords: Acromegaly; Pegvisomant; Osteoporosis
MeSH Terms: conditions — Acromegaly; Osteoporosis | interventions — pegvisomant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Peripheral blood specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Acromegaly patients on pegvisomant: 25 subjects with acromegaly on pegvisomant therapy with a normal IGF-1 level for at least 1 year.
  Interventions: Drug: Pegvisomant

INTERVENTIONS:
Drug: Pegvisomant — Subjects receiving pegvisomant as part of their clinical care for acromegaly will be studied.
  Other Names: Somavert

SUMMARY:
The investigators will conduct a cross-sectional study of bone density, bone microarchitecture, vertebral fractures and trabecular bone score in 25 patients with acromegaly treated with Pegvisomant, the growth hormone (GH) receptor antagonist for at least 1 year and with normal insulin-like growth factor-1 (IGF-1) levels. This study aims to describe the bone architecture and associated biochemical indices of bone turnover and metabolism in patients with active acromegaly and how these are altered with treatment of the disease.

DETAILED DESCRIPTION:
Growth hormone (GH) and Insulin-Like Growth Factor-1 (IGF-1) are important regulators of bone modeling and remodeling, fundamental to maintenance of normal skeletal integrity. In acromegaly, a disease characterized by longstanding exposure to excess GH and IGF-1, these hormones induce marked skeletal changes. Most dual energy X-ray absorptiometry (DXA) studies report that bone mineral density (BMD) is normal in acromegaly. Despite this, however, there is mounting evidence that bone health is adversely affected in patients with both active and successfully treated acromegaly.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with acromegaly
* On pegvisomant therapy with a normal IGF-1 level for at least 1 year

Exclusion Criteria:

* Malignancy (except cured basal, squamous cell skin carcinoma or other cured cancers free from recurrence > 3 years)
* Pregnancy or lactation within last 12 months
* Untreated primary hyperparathyroidism, hyper- or hypothyroidism
* Cushing's syndrome
* Prolactin-secreting pituitary adenoma
* GH deficiency
* On current drug therapy for osteoporosis
* Diabetes mellitus
* Renal insufficiency
* Liver disease
* Current or past use of glucocorticoids (more than physiologic dose), anticonvulsants, anticoagulants, methotrexate, aromatase inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 25 subjects with acromegaly on pegvisomant therapy with a normal IGF-1 level for at least 1 year will be studied.
  Patients will be on stable doses of any pituitary hormone supplements for 3 months prior to study entry including gonadal steroid replacement for men or premenopausal women. Hypogonadal men and premenopausal women will be replaced with clinically appropriate sex steroid replacement. Subjects will be 50% females.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2016-08-03 (Actual); Primary Completion 2019-12-21 (Actual); Study Completion 2019-12-21 (Actual)

PRIMARY OUTCOMES:
Volumetric bone mineral density of radius (vBMD) | Measured once at one study visit
  Volumetric bone mineral density of radius (vBMD) measured by high resolution peripheral quantitative computed tomography (HRpQCT)

SECONDARY OUTCOMES:
Trabecular number of radius (TbN) | Measured once at one study visit
  HRpQCT determined bone microarchitecture
Trabecular Thickness of radius (Tb.Th) | Measured once at one study visit
  HRpQCT determined bone microarchitecture
Trabecular separation of radius (Tb.Sp) | Measured once at one study visit
  HRpQCT determined bone microarchitecture
Cortical density of radius | Measured once at one study visit
  HRpQCT determined bone microarchitecture
Cortical thickness of radius | Measured once at one study visit
  HRpQCT determined bone microarchitecture
Areal bone mineral density (aBMD) of lumbar sacral spine | Measured once at one study visit
  Areal bone mineral density of lumbar sacral spine determined by DXA
Trabecular bone score of LS spine | Measured once at one study visit
  Trabecular bone score of lumbar sacral (LS) spine determined by DXA

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Freda, MD, Principal Investigator — Columbia University
Locations (1):
- Neuroendocrine Unit and Pituitary Center, Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided